CLINICAL TRIAL: NCT06601504
Title: A Phase II Randomized, Controlled Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of HMPL-760 Plus R-GemOx Versus Placebo Plus R-GemOx in Patients With Relapsed/Refractory Diffuse Large B-Cell Lymphoma(R/R DLBCL)
Brief Title: Study of HMPL-760 Plus R-GemOx Versus Placebo Plus R-GemOx in Relapsed/Refractory DLBCL
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hutchmed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-760-00CH1
Record Dates: First submitted 2024-09-08; First posted 2024-09-19 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Relapsed/Refractory Diffuse Large B-Cell Lymphoma
Keywords: R-GemOx; R/R DLBCL; HMPL-760
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab; Gemcitabine; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A: HMPL-760 planned dose 1 once daily (QD) in combination with R-GemOx regimen (Experimental): Group A: Patients will receive HMPL-760 planned dose 1 once daily (QD) orally from Cycle 1 Day 1 until disease progression(PD), patient death, intolerable toxicity, etc., in combination with R-GemOx regimen in 21-day cycle for a total of 6 cycles. Rituximab 375 mg/m^2 ivgtt is given on day 1 of each cycle, and gemcitabine 1000 mg/m^2 ivgtt is given, followed by oxaliplatin 100 mg/m^2 ivgtt on day 2 of each cycle.
  Interventions: Drug: HMPL-760 planned dose 1; Drug: R-GemOx
- Group B: HMPL-760 placebo planned dose 1 once daily (QD) in combination with R-GemOx regimen (Placebo Comparator): Patients will receive HMPL-760 placebo planned dose 1 once daily (QD) orally from Cycle 1 Day 1 until disease progression(PD), patient death, intolerable toxicity, etc., in combination with R-GemOx regimen in 21-day cycle for a total of 6 cycles. Rituximab 375 mg/m^2 ivgtt is given on day 1 of each cycle, and gemcitabine 1000 mg/m^2 ivgtt is given, followed by oxaliplatin 100 mg/m^2 ivgtt on day 2 of each cycle.
  Interventions: Drug: R-GemOx; Drug: HMPL-760 placebo planned dose 1
- Group C: HMPL-760 planned dose 2 once daily (QD) in combination with R-GemOx regimen (Experimental): Patients will receive HMPL-760 planned dose 2 once daily (QD) orally from Cycle 1 Day 1 until disease progression(PD), patient death, intolerable toxicity, etc., in combination with R-GemOx regimen in 21-day cycle for a total of 6 cycles. Rituximab 375 mg/m^2 ivgtt is given on day 1 of each cycle, and gemcitabine 1000 mg/m^2 ivgtt is given, followed by oxaliplatin 100 mg/m^2 ivgtt on day 2 of each cycle.
  Interventions: Drug: R-GemOx; Drug: HMPL-760 planned dose 2
- Group D: HMPL-760 placebo planned dose 2 once daily (QD) in combination with R-GemOx regimen (Placebo Comparator): Patients will receive HMPL-760 placebo planned dose 2 once daily (QD) orally from Cycle 1 Day 1 until disease progression(PD), patient death, intolerable toxicity, etc., in combination with R-GemOx regimen in 21-day cycle for a total of 6 cycles. Rituximab 375 mg/m^2 ivgtt is given on day 1 of each cycle, and gemcitabine 1000 mg/m^2 ivgtt is given, followed by oxaliplatin 100 mg/m^2 ivgtt on day 2 of each cycle.
  Interventions: Drug: R-GemOx; Drug: HMPL-760 placebo planned dose 2

INTERVENTIONS:
Drug: HMPL-760 planned dose 1 — HMPL-760 planned dose 1 daily (QD) orally
  Arms: Group A: HMPL-760 planned dose 1 once daily (QD) in combination with R-GemOx regimen
Drug: R-GemOx — R-GemOx regimen includes Rituximab Injection, Gemcitabine Hydrochloride for Injection, Gemcitabine Hydrochloride for Injection. R-GemOx regimen in 21-day cycle for a total of 6 cycles. Rituximab 375 mg/m^2 ivgtt is given on day 1 of each cycle, and gemcitabine 1000 mg/m^2 ivgtt is given, followed by oxaliplatin 100 mg/m^2 ivgtt on day 2 of each cycle.
  Other Names: Rituximab Injection, Gemcitabine Hydrochloride for Injection, Gemcitabine Hydrochloride for Injection
Drug: HMPL-760 placebo planned dose 1 — HMPL-760 placebo planned dose 1 daily (QD) orally
  Arms: Group B: HMPL-760 placebo planned dose 1 once daily (QD) in combination with R-GemOx regimen
Drug: HMPL-760 planned dose 2 — HMPL-760 planned dose 2 daily (QD) orally
  Arms: Group C: HMPL-760 planned dose 2 once daily (QD) in combination with R-GemOx regimen
Drug: HMPL-760 placebo planned dose 2 — HMPL-760 placebo planned dose 2 daily (QD) orally
  Arms: Group D: HMPL-760 placebo planned dose 2 once daily (QD) in combination with R-GemOx regimen

SUMMARY:
The goal of this study is to evaluate the efficacy of HMPL-760 in combination with R-GemOx versus placebo in combination with R-GemOx in patients with Relapsed/Refractory Diffuse Large B-Cell Lymphoma (R/R DLBCL).

DETAILED DESCRIPTION:
A Phase II Randomized, Controlled Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of HMPL-760 in Combination with R-GemOx versus Placebo in Combination with R-GemOx in Patients with Relapsed/Refractory Diffuse Large B-Cell Lymphoma (R/R DLBCL). The study phases include screening period, treatment period, safety observation period, PFS follow-up period, and OS follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the Informed consent form(ICF) and be able to follow the requirements of study protocol;
2. Age ≥18 years;
3. Eastern Cooperative Oncology Group (ECOG) performance status between 0 and 2;
4. Histopathologically confirmed diagnosis of DLBCL;
5. The investigator judges that the patient's current condition requires further treatment;
6. Patients should have at least one bi-dimensionally measurable lesion;
7. Expected survival is more than 12 weeks;

Exclusion Criteria:

1. Patients with known primary or secondary central nervous system lymphoma (CNSL) or the presence of clinical symptoms suggestive of CNSL;
2. Women who are pregnant (positive pregnancy test during the screening period) or breastfeeding;
3. Organ insufficiency;
4. Currently known history of liver disease, including cirrhosis, alcoholic liver, known active infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV):
5. History of significant organ bleeding, including gastrointestinal bleeding, hematencephalon, haemoptysis, etc., within 8 weeks prior to the first dose of study drug;
6. Known risk of bleeding, such as coagulation factor deficiency, vascular hemophilia; or the patient is receiving vitamin K antagonist (warfarin);
7. Toxicities from prior anticancer therapy not resolved to Grade ≤ 1 (except for alopecia and decreased appetite);
8. Clinically significant active infection;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2024-11-05 (Actual); Primary Completion 2026-05-12 (Estimated); Study Completion 2026-11-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Up to approximately 2 years
  Progression-free survival (PFS): Efficacy is evaluated using the Lugano Efficacy Evaluation Criteria for Malignant Lymphoma (Cheson 2014).

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 2 years
  Objective Response Rate (ORR) is defined as the ratio of patients who reached complete response (CR) or partial response (PR), as assessed by investigator.
Complete response (CR) rate | Up to approximately 2 years
  Complete response (CR) rate is defined as the ratio of patients with who reached complete response (CR), as assessed by investigator.
Duration of response (DoR) | Up to approximately 2 years
  For patients who reached complete response (CR) or partial response (PR), Duration of Response (DoR) is defined as the time from the first CR or PR until disease progression or death due to any cause, whichever occurs first, as assessed by investigator.
Clinical benefit rate (CBR) | Up to approximately 2 years
  Defined as the ratio of patients with complete response (CR), partial response (PR), or stable disease (SD).
Time to response (TTR) | Up to approximately 2 years
  Time To Response (TTR) is defined as the time from the start of treatment to the first objective response rate (ORR), as assessed by investigator.
Overall survival (OS) | Up to approximately 2 years
  Overall Survival (OS) is defined as the time from randomization to death due to any cause.
Safety Endpoints of adverse events | Up to approximately 2 years
  Incidence and severity of treatment-emergent adverse events (TEAEs), incidence of serious adverse events (SAEs), incidence of TEAEs leading to permanent discontinuation, dose interruption, and dose reduction, and their correlation to study drug. The severity is determined according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 (NCI CTCAE 5.0).
Pharmacokinetic(PK) profile of HMPL-760 in combination with R-GemOx | At the end of Cycle 7 (each cycle is 21 days)
  Trough plasma concentration (Ctrough) of drug
Pharmacokinetic(PK) profile of HMPL-760 in combination with R-GemOx | At the end of Cycle 7 (each cycle is 21 days)
  Maximum observed concentration, occurring at time Tmax at steady-state (Cmax,ss) of drug
Pharmacokinetic(PK) profile of HMPL-760 in combination with R-GemOx | At the end of Cycle 7 (each cycle is 21 days)
  Time of maximum observed concentration at steady-state(Tmax,ss) of drug
Pharmacokinetic(PK) profile of HMPL-760 in combination with R-GemOx | At the end of Cycle 7 (each cycle is 21 days)
  The partial area from dosing time to dosing time plus Tau at steady-state (AUCss) of drug
Pharmacokinetic(PK) profile of HMPL-760 in combination with R-GemOx | At the end of Cycle 7 (each cycle is 21 days)
  Apparent clearance at steady-state (CLss/F) of drug (if applicable)
Pharmacokinetic(PK) profile of HMPL-760 in combination with R-GemOx | At the end of Cycle 7 (each cycle is 21 days)
  Apparent volume of distribution at steady-state (Vz,ss/F) of drug (if applicable)

OTHER OUTCOMES:
Biomarker assessment | Up to approximately 2 years
  To evaluate the correlation between potential biomarkers and the prognosis of patients treated with this regimen. Tumor tissue or blood samples will be examined to detect the gene expression of MYD88.
Metabolite analysis of HMPL-760 in combination with R-GemOx | At the end of Cycle 7 (each cycle is 21 days)
  Analysis metabolite of HMPL-760 in combination with R-GemOx

CONTACTS AND LOCATIONS:
Overall Officials: Weili Zhao, Principal Investigator — Ruijin Hospital
Locations (16):
- China (16):
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Guangxi Medical University Cancer Hospital, Nanning, Guangxi
  - Wuhan Union Hospital of China, Wuhan, Hebei
  - Harbin First Hospital, Harbin, Heilongjiang
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Jiangxi Cancer Hospital, Nanchang, Jiangxi
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Shandong Cancer Hospital & Institute, Jinan, Shandong
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No